CLINICAL TRIAL: NCT03634488
Title: Management of Severe Acute Malnutrition in Children With Sickle Cell Disease Greater Than 5 Years of Age Living in Northern Nigeria
Brief Title: Management of Severe Acute Malnutrition in SCD, in Northern Nigeria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Aminu Kano Teaching Hospital (Other); Murtala Muhammad Specialist Hospital (Other)
Responsible Party: Principal Investigator, Michael DeBaun, Vice Chair for Clinical Research, JC Peterson Endowed Chair, Professor of Pediatrics and Medicine, Director, Vanderbilt-Meharry-Matthew Walker Center of Excellence in Sickle Cell Disease, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 170577
Record Dates: First submitted 2018-01-30; First posted 2018-08-16 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-02

CONDITIONS: Sickle Cell Anemia; Severe Acute Malnutrition
Keywords: sickle cell disease; sub-Saharan Africa; malnutrition; low-income settings; severe acute malnutrition; sickle cell anemia; Nigeria
MeSH Terms: conditions — Anemia, Sickle Cell; Severe Acute Malnutrition; Malnutrition | interventions — Hydroxyurea

STUDY DESIGN:
Intervention Model Description: A 12-week, open label, randomized controlled feasibility trial in children with sickle cell anemia between 5 and 12 years of age to treat uncomplicated severe malnutrition.
Who Masked: Investigator
Masking Description: Allocation was concealed from all other study personnel, except statisticians.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- SCD - Ready-to-use therapeutic food and Hydroxyurea (Experimental): 50-75 children (5-12 years old) with SCA and severe malnutrition will be randomly allocated to receive ready-to-use therapeutic food and hydroxyurea (20mg/kg/day)
  Interventions: Drug: hydroxyurea (20mg/kg/day); Dietary Supplement: Ready-to-use therapeutic food
- SCD - Ready-to-use therapeutic food alone (Placebo Comparator): 50-75 children (5-12 years old) with SCA and severe malnutrition will be randomly allocated to receive ready-to-use therapeutic food alone
  Interventions: Dietary Supplement: Ready-to-use therapeutic food
- Non-SCD siblings with severe malnutrition (Placebo Comparator): To decrease the likelihood of sharing limited food resources, we will enroll up to 100 malnourished non-SCD siblings.
  Interventions: Dietary Supplement: Ready-to-use therapeutic food

INTERVENTIONS:
Drug: hydroxyurea (20mg/kg/day) — Treatment of severe malnutrition in children with SCA in northern Nigeria
  Other Names: hydrea
  Arms: SCD - Ready-to-use therapeutic food and Hydroxyurea
Dietary Supplement: Ready-to-use therapeutic food — Treatment of severe malnutrition in children with and without SCA in northern Nigeria with an additional 500-1000 calories from ready-to-use-therapeutic food
  Other Names: RUTF

SUMMARY:
Except for children with HIV, all recommendations for treatment of childhood malnutrition are for children < 5 years of age. The overall goal of this randomized controlled nutrition feasibility trial is to identify whether families of children with sickle cell disease (SCD) 5 years and older agree to participate over a 12-week period. The investigators will also establish a safety protocol for monitoring potential complications associated with treating severe malnutrition in children 5 years and older with and without SCD, in a low-resource setting.

DETAILED DESCRIPTION:
The overall goal of this feasibility trial is to determine the acceptability of a randomized controlled trial to ascertain the optimal strategy for the treatment of severe malnutrition in children with sickle cell disease (SCD) 5 years and older. No international standard or evidence-based guidelines exist for the treatment of severe malnutrition (defined as BMI Z-score below -3) in children with SCD. With an expanding pediatric population of more than 75 million in Nigeria, coupled with decreasing childhood infectious disease-related mortality, the next emerging threats to preventable childhood deaths are non-communicable diseases. Data from our NIH-funded randomized controlled primary stroke prevention trial in Nigeria (NCT02560935), in which the investigators evaluated children with SCD between 5 and 12 years of age, demonstrated that 29% (230/803) of the cohort met criteria for severe malnutrition. Approximately 92% of the cohort in northern Nigeria identified as having severe malnutrition was below the 5th percentile for weight of children with SCD living in the US, Canada, or Europe. These data indicate older children with SCD living in northern Nigeria are undernourished when compared to children living with SCD in high-resource settings. A potentially unique attribute to treating malnutrition in children with SCD is the use of FDA approved anti-metabolite, hydroxyurea, to prevent vaso-occlusive pain events in children. The beneficial effects of hydroxyurea include, but are not limited to, decreased inflammation and increased hemoglobin levels. Preliminary evidence in this cohort of older children with sickle cell anemia (SCA) in northern Nigeria reveals that moderate fixed-dose hydroxyurea (20 mg/kg/day) significantly increases BMI in children with severe malnutrition. The investigators propose a randomized controlled feasibility trial in older children (5 to 12 years of age) with SCA living in northern Nigeria. In preparation for a definitive phase III trial to determine if ready-to-use therapeutic food and moderate fixed-dose hydroxyurea therapy is superior to ready-to-use therapeutic food alone, the investigators will randomly allocate up to 150 children between 5 and 12 years of age with SCA and severe uncomplicated malnutrition to each of the two arms. In aim 1, the investigators will assess the feasibility (rate of recruitment, retention, and adherence) of a randomized controlled trial (RCT) in children with SCD and severe malnutrition to a 12-week intervention period. For aim 2, the investigators will establish the safety protocol to monitor for unknown rates of complications associated with treating malnutrition in children with SCD. To decrease the likelihood of sharing limited food resources in a poor family and to determine the specificity of malnutrition for children with SCD in northern Nigeria, the investigators will screen and treat up to 100 malnourished non-SCD siblings of the trial participants. After completion of this feasibility trial, the investigators will use the acquired knowledge to design a phase III trial to definitively determine the optimal treatment strategy for severe malnutrition in older children with SCD living in Africa, potentially affecting thousands of children in this region.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnoses of SCA, comparison children without SCD
* severe malnutrition defined as a BMI z-score < -3
* age between 5 and 12 years (assessment can take place up until the 13th birthday)
* pass the appetite test
* uncomplicated malnutrition (good appetite, alert, no signs of infection of respiratory distress)

Exclusion Criteria:

* children with complicated severe acute malnutrition
* children with electrolyte disturbances (serum Na, K, PO4) at baseline
* children on disease-modifying therapy (hydroxyurea or regular blood transfusion therapy)
* children enrolled in other studies
* children with diabetes and other chronic illnesses
* children with known HIV infection
* children with a known allergy to dairy or peanuts.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 132 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael DeBaun, Principal Investigator — Vanderbilt University Medical Center
Locations (3):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States
- Nigeria (2):
  - Aminu Kano Teaching Hospital, Kano
  - Murtala Mohammad Specialist Hospital, Kano

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murtala HA, Abdullahi SU, Gambo S, Kabir H, Shamsu KA, Gwarzo G, Acra SA, Stallings VA, Rodeghier M, DeBaun MR, Klein LJ. Including malnourished siblings in treatment improves nutritional outcomes for children with sickle cell anemia in Northern Nigeria: Results from a feasibility trial. Nutr Res. 2025 Dec;144:32-37. doi: 10.1016/j.nutres.2025.10.006. Epub 2025 Oct 18. PMID 41253090
- [Derived] Brechko A, Abdullahi SU, Gambo S, Murtala HA, Kabir H, Shamsu KA, Stallings VA, Rodeghier M, Ramesh A, Sellers A, Schlundt DG, DeBaun MR, Klein LJ. Adherence to ready-to-use therapeutic food in older children with sickle cell anaemia and severe acute malnutrition: a mixed-methods study in a low-income setting. BMJ Glob Health. 2025 Aug 7;10(8):e019096. doi: 10.1136/bmjgh-2025-019096. PMID 40780831
- [Derived] Ramirez-Cuebas G, Abdullahi SU, Gambo S, Murtala HA, Kabir H, Shamsu KA, Gwarzo G, Acra SA, Stallings VA, Rodeghier M, DeBaun MR, Klein LJ. Impact of Food Insecurity on Malnutrition Treatment Response in Nigerian Children With Sickle Cell Anemia and Severe Acute Malnutrition. Pediatr Blood Cancer. 2025 Jun;72(6):e31637. doi: 10.1002/pbc.31637. Epub 2025 Mar 10. PMID 40062628
- [Derived] Ritter C, Abdullahi SU, Gambo S, Murtala HA, Kabir H, Shamsu KA, Gwarzo G, Banaei Y, Acra SA, Stallings VA, Rodeghier M, DeBaun MR, Klein LJ. Impact of maternal depression on malnutrition treatment outcomes in older children with sickle cell anemia. BMC Nutr. 2024 Jan 24;10(1):18. doi: 10.1186/s40795-024-00826-0. PMID 38268013
- [Derived] Abdullahi SU, Gambo S, Murtala HA, Kabir H, Shamsu KA, Gwarzo G, Acra S, Stallings VA, Rodeghier M, DeBaun MR, Klein LJ. Feasibility trial for the management of severe acute malnutrition in older children with sickle cell anemia in Nigeria. Blood Adv. 2023 Oct 24;7(20):6024-6034. doi: 10.1182/bloodadvances.2023010789. PMID 37428866

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was enrolled in the "Management of Severe Acute Malnutrition in Children With Sickle Cell Disease Greater Than 5 Years of Age Living in Northern Nigeria" study in August 2021. Recruitment took place at Aminu Kano Teaching Hospital and Murtala Muhammad Specialist Hospital in Kano, Nigeria. Enrollment for children with SCD (either the Ready-to-Use Therapeutic Food arm or the Ready-to-Use Therapeutic Food and Hydroxyurea arm) and siblings without SCD ended in May 2022.
Pre-assignment Details: The feasibility trial's primary objectives are to evaluate the intervention's feasibility and safety in children with sickle cell anemia.
Groups:
- SCD: Ready-to-use Therapeutic Food and Hydroxyurea: At least 50 children (5-12 years old) with SCA and severe malnutrition will be randomly allocated to receive Ready-to-use therapeutic food (500-1,000 daily calories) and hydroxyurea (20mg/kg/day)
  Hydroxyurea (20mg/kg/day): Treatment of severe malnutrition in children with SCA in northern Nigeria
  Ready-to-use therapeutic food: Treatment of severe malnutrition in children with SCA in northern Nigeria with an additional 500-1000 calories from ready-to-use-therapeutic food
- SCD: Ready-to-use Therapeutic Food Alone: At least 50 children (5-12 years old) with SCA and severe malnutrition will be randomly allocated to receive Ready-to-use therapeutic food alone
  Ready-to-use therapeutic food: Treatment of severe malnutrition in children with SCA in northern Nigeria with an additional 500-1000 calories from ready-to-use-therapeutic food
- Siblings Without SCD: Up to 100 non-SCD siblings(5-12 years old) and severe malnutrition will be enrolled.
  Ready-to-use therapeutic food: Treatment of severe malnutrition in children without SCD in northern Nigeria with an additional 500-1000 calories from ready-to-use-therapeutic food
Period: Overall Study
Arm/Group | SCD: Ready-to-use Therapeutic Food and Hydroxyurea | SCD: Ready-to-use Therapeutic Food Alone | Siblings Without SCD
Started | 56 | 54 | 22
Completed | 54 | 54 | 22
Not Completed | 2 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — A participant was administratively withdrawn due to a calculated BMI z-score >-3.0. | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics of participants with sickle cell anemia and severe acute malnutrition by randomization status in the SAMS trial. Baseline characteristics of non-SCD siblings with sickle cell anemia and severe acute malnutrition by randomization status in the SAMS trial.
Groups:
- SCD - Ready-to-use Therapeutic Food and Hydroxyurea: Children (5-12 years old) with SCA and severe malnutrition randomly allocated to receive Ready-to-use therapeutic food and hydroxyurea (20mg/kg/day)
  hydroxyurea (20mg/kg/day): Treatment of severe malnutrition in children with SCA in northern Nigeria
  Ready-to-use therapeutic food: Treatment of severe malnutrition in children with SCA in northern Nigeria with an additional 500-1000 calories from ready-to-use-therapeutic food
- SCD - Ready-to-use Therapeutic Food Alone: Children (5-12 years old) with SCA and severe malnutrition randomly allocated to receive Ready-to-use therapeutic food alone
  Ready-to-use therapeutic food: Treatment of severe malnutrition in children with SCA in northern Nigeria with an additional 500-1000 calories from ready-to-use-therapeutic food
- Siblings Without SCD: non-SCD siblings(5-12 years old) with severe malnutrition.
  Ready-to-use therapeutic food: Treatment of severe malnutrition in children without SCD in northern Nigeria with an additional 500-1000 calories from ready-to-use-therapeutic food
- Total: Total of all reporting groups
Arm/Group | SCD - Ready-to-use Therapeutic Food and Hydroxyurea | SCD - Ready-to-use Therapeutic Food Alone | Siblings Without SCD | Total
Number analyzed (Participants) | 55 | 54 | 22 | 131
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 10.2 [8.2 to 11.4] | 10.5 [9.4 to 11.7] | 8.2 [7.0 to 10.7] | 10.1 [8.2 to 11.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 27 | 14 | 67
  Male | 29 | 27 | 8 | 64
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Fulani | 4 | 2 | 0 | 6
  Hausa | 49 | 51 | 22 | 122
  Kanuri | 1 | 0 | 0 | 1
  Other | 1 | 1 | 0 | 2
Weight, kg, mean (std. dev.) [Mean (Standard Deviation); unit: kg] | 18.4 (3.5) | 18.7 (3.5) | 18.1 (4.2) | 18.5 (3.6)
Height, cm, mean (std. dev.) [Mean (Standard Deviation); unit: centimeters] | 123.5 (10.1) | 124.1 (9.5) | 123.5 (12.3) | 123.7 (10.2)
Body Mass Index, kg/m^2, mean (std. dev.) [Mean (Standard Deviation); unit: kg/m^2] | 12 (0.6) | 12.1 (0.6) | 11.7 (0.6) | 12 (0.6)
Body Mass Index z-score, mean (std. dev.) [Mean (Standard Deviation); unit: Z-score] — Using the World Health Organization (WHO) growth reference, anthropometric measurements were converted to age and sex-specific z-scores. Anthropometric Indices (BMI-for-age (BMIZ), were calculated using WHO 2007 R Macro Package to assess growth and development of the children. Severe malnutrition/wasting (SAM) was defined as a body mass index (BMI) z-score <-3.0.
  Z-score | -3.64 (0.49) | -3.66 (0.44) | -3.6 (0.5) | -3.65 (0.46)
Hemoglobin, g/dl, mean (std. dev.) [Mean (Standard Deviation); unit: g/dl] | 7.4 (1) | 7.3 (1.1) | 10.8 (1.0) | 7.9 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Enrollment Rate at the End of the 6-month Recruitment Period
Description: Recruitment Feasibility: The primary outcome is the proportion of eligible individuals that agree to be included, referred to as the recruitment rate. Children with severe malnutrition who qualified and agreed to participate were invited to sign a consent and assent for study recruitment to this study.
Time Frame: 6 months
Population: Children aged 5-12 years with SCA were evaluated for eligibility. Siblings of enrolled participants aged 5-12 years old without SCD were also evaluated for eligibility.
Measure: Number; unit: participants
Groups:
- Eligible Children Aged 5-12 Years With SCA: Children with SCA who met the criteria to participate in the study
- Eligible Children Aged 5-12 Years Old Without SCD: Non-SCD siblings of participants with SCA who met the criteria to participate in the study
Arm/Group | Eligible Children Aged 5-12 Years With SCA | Eligible Children Aged 5-12 Years Old Without SCD
Number analyzed (Participants) | 111 | 22
participants
  Eligible | 111 | 22
  Randomized | 110 | 22
  Unable to randomize | 1 | 0

2. Primary Outcome: Retention Over 12-week Period
Description: The primary outcome is the proportion of participants who completed the 12-week trial, known as the retention rate for the trial.
Time Frame: 12 weeks
Population: The analysis included participants with sickle cell anemia and severe acute malnutrition. The feasibility trial's primary objectives are to evaluate the intervention's feasibility and safety in children with sickle cell anemia.
Measure: Number; unit: participants
Groups:
- SCD - Ready-to-use Therapeutic Food and Hydroxyurea: Children (5-12 years old) with SCA and severe malnutrition were randomly allocated to receive Ready-to-use therapeutic food (500-1,000 daily calories) and hydroxyurea (20mg/kg/day)
- SCD - Ready-to-use Therapeutic Food Alone: Children (5-12 years old) with SCA and severe malnutrition randomly allocated to receive Ready-to-use therapeutic food (500-1,000 daily calories) only.
- Siblings Without SCD: Non-SCD siblings (5-12 years old) with severe malnutrition enrolled to receive Ready-to-use therapeutic food (500-1,000 daily calories) only.
Arm/Group | SCD - Ready-to-use Therapeutic Food and Hydroxyurea | SCD - Ready-to-use Therapeutic Food Alone | Siblings Without SCD
Number analyzed (Participants) | 56 | 54 | 22
participants
  Voluntarily withdrew from the trial | 0 | 0 | 0
  Involuntary withdrawal from the trial | 1 | 0 | 0

3. Primary Outcome: Percentage of Ready-to-use Therapeutic Food Sachets Returned as Empty.
Description: Adherence to the ready-to-use therapeutic food was evaluated based on the percentage of empty food sachets returned at each visit.
Time Frame: 12 weeks
Population: The final analysis included 54 participants with sickle cell anemia from each arm with sickle cell anemia and severe acute malnutrition, along with 22 non-SCD siblings with severe acute malnutrition.
Measure: Mean (95% Confidence Interval); unit: percentage of empty sachets
Groups:
- SCD - Ready-to-use Therapeutic Food Alone: Children (5-12 years old) with SCA and severe malnutrition were randomly allocated to receive Ready-to-use therapeutic food (500-1,000 daily calories) only.
Arm/Group | SCD - Ready-to-use Therapeutic Food and Hydroxyurea | SCD - Ready-to-use Therapeutic Food Alone | Siblings Without SCD
Number analyzed (Participants) | 54 | 54 | 22
percentage of empty sachets | 99.02 [99.00 to 99.04] | 99.03 [99.0 to 99.05] | 99.02 [99.01 to 99.04]

4. Primary Outcome: Number of Missed Visits
Description: Adherence to monthly visits was assessed based on the number of missed visits
Time Frame: 12 weeks
Population: Per-protocol analysis of participants.
Measure: Number; unit: missed visits
Units Other Than Participants: Research Visits
Arm/Group | SCD - Ready-to-use Therapeutic Food and Hydroxyurea | SCD - Ready-to-use Therapeutic Food Alone | Siblings Without SCD
Number analyzed (Participants) | 54 | 54 | 22
Number analyzed (Research Visits) | 216 | 216 | 88
missed visits | 0 | 0 | 0

5. Primary Outcome: Percentage of Hydroxyurea Pills Returned
Description: Adherence to hydroxyurea was evaluated based on the percentage of hydroxyurea pills returned for the group randomized to both ready-to-use therapeutic food and hydroxyurea.
Time Frame: 12 weeks
Population: The final analysis included 54 participants with sickle cell anemia and severe acute malnutrition randomized to receive hydroxyurea in addition to ready-to-use therapeutic food. The other arms did not receive hydroxyurea, and therefore, adherence to hydroxyurea cannot be evaluated.
Measure: Mean (95% Confidence Interval); unit: percentage of hydroxyurea pills returned
Arm/Group | SCD - Ready-to-use Therapeutic Food and Hydroxyurea
Number analyzed (Participants) | 54
percentage of hydroxyurea pills returned | 4.4 [0.00 to 8.27]

6. Primary Outcome: Change in Mean Corpuscular Volume
Description: Adherence to hydroxyurea was evaluated based on change in mean corpuscular volume
Time Frame: 12 weeks
Population: The final analysis included 54 participants from each arm with sickle cell anemia and severe acute malnutrition. We did not include the siblings' change in mean corpuscular volume - since none of the siblings without sickle cell disease received hydroxyurea.
Measure: Mean (Standard Deviation); unit: fl
Groups:
- Ready-to-use Therapeutic Food and Hydroxyurea: Children (5-12 years old) with SCA and severe malnutrition were randomly allocated to receive Ready-to-use therapeutic food (500-1,000 daily calories) and hydroxyurea (20mg/kg/day).
- Ready-to-use Therapeutic Food Alone: Children (5-12 years old) with SCA and severe malnutrition were randomly allocated to receive Ready-to-use therapeutic food (500-1,000 daily calories).
Arm/Group | Ready-to-use Therapeutic Food and Hydroxyurea | Ready-to-use Therapeutic Food Alone
Number analyzed (Participants) | 54 | 54
fl | 5.4 (12.7) | -1.0 (10.9)

7. Primary Outcome: Change in Fetal Hemoglobin Level Percentage
Description: The primary outcome is the proportion of eligible individuals who adhere to therapy (Ready-to-use therapeutic food and hydroxyurea). The adherence rate for hydroxyurea was determined based on the change in fetal hemoglobin level percentage.
Time Frame: Baseline to 12 weeks
Population: The final analysis included 54 participants from each arm with sickle cell anemia and severe acute malnutrition. We did not measure fetal hemoglobin in children without SCD.
Measure: Median (Inter-Quartile Range); unit: percentage of fetal hemoglobin
Groups:
- Ready-to-use Therapeutic Food Alone: Children (5-12 years old) with SCA and severe malnutrition were randomly allocated to receive Ready-to-use therapeutic food (500-1,000 daily calories) only.
Arm/Group | SCD - Ready-to-use Therapeutic Food and Hydroxyurea | Ready-to-use Therapeutic Food Alone
Number analyzed (Participants) | 54 | 54
percentage of fetal hemoglobin | 3.9 [1.7 to 6.8] | 2.2 [0.5 to 4.9]

8. Primary Outcome: Mean Corpuscular Volume Values at Exit
Description: The primary outcome is the proportion of eligible individuals who adhere to therapy (Ready-to-use therapeutic food and hydroxyurea). The adherence rate for hydroxyurea was determined based on mean corpuscular volume (MCV) values at exit (12 weeks).
Time Frame: Feasibility over 12-week Period [Time Frame: 3 months]
Population: The final analysis included 54 participants from each arm with sickle cell anemia and severe acute malnutrition. The feasibility trial's primary objectives are to evaluate the intervention's feasibility and safety in children with sickle cell anemia. We, therefore, did not include the outcomes for the siblings in these main results.
Measure: Mean (Standard Deviation); unit: fl
Groups:
- Ready-to-use Therapeutic Food and Hydroxyurea: At least 50 children (5-12 years old) with SCA and severe malnutrition will be randomly allocated to receive Ready-to-use therapeutic food and hydroxyurea (20mg/kg/day)
  hydroxyurea (20mg/kg/day): Treatment of severe malnutrition in children with SCA in northern Nigeria
  Ready-to-use therapeutic food: Treatment of severe malnutrition in children with SCA in northern Nigeria with an additional 500-1000 calories from ready-to-use-therapeutic food
- Ready-to-use Therapeutic Food Alone: At least 50 children (5-12 years old) with SCA and severe malnutrition will be randomly allocated to receive Ready-to-use therapeutic food alone
  Ready-to-use therapeutic food: Treatment of severe malnutrition in children with SCA in northern Nigeria with an additional 500-1000 calories from ready-to-use-therapeutic food
Arm/Group | Ready-to-use Therapeutic Food and Hydroxyurea | Ready-to-use Therapeutic Food Alone
Number analyzed (Participants) | 54 | 54
fl | 88.5 (14.7) | 85.4 (11.4)

9. Primary Outcome: Fetal Hemoglobin Levels at Exit
Description: The primary outcome is the proportion of eligible individuals who adhere to therapy (Ready-to-use therapeutic food and hydroxyurea). The adherence rate for hydroxyurea was determined based on the fetal hemoglobin levels at exit (12 weeks).
Time Frame: Feasibility over 12-week Period [Time Frame: 3 months]
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: percentage of fetal hemoglobin
Arm/Group | Ready-to-use Therapeutic Food and Hydroxyurea | Ready-to-use Therapeutic Food Alone
Number analyzed (Participants) | 54 | 54
percentage of fetal hemoglobin | 12.2 [7.5 to 16.9] | 9.4 [5.6 to 13.8]

10. Primary Outcome: Total Hemoglobin Levels at Exit
Description: The primary outcome is the proportion of eligible individuals who adhere to therapy (Ready-to-use therapeutic food and hydroxyurea). The adherence rate for hydroxyurea was determined based on the total hemoglobin levels at exit (12 weeks).
Time Frame: Feasibility over 12-week Period [Time Frame: 3 months]
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Ready-to-use Therapeutic Food and Hydroxyurea | Ready-to-use Therapeutic Food Alone
Number analyzed (Participants) | 54 | 54
g/dl | 8.3 (1.1) | 7.7 (1.3)

11. Secondary Outcome: Percentage of Participants Maintaining a BMI Z-score Less Than -3.0
Description: As a secondary outcome, we assessed the percentage of participants with and without SCA who continued to have a body mass index z-score of <-3.0 at the end of the 12 weeks of treatment. Using the World Health Organization (WHO) growth reference, anthropometric measurements were converted to age and sex-specific z-scores. Anthropometric Indices (BMI-for-age (BMIZ), were calculated using WHO 2007 R Macro Package to assess growth and development of the children. Severe malnutrition/wasting (SAM) was defined as a body mass index (BMI) z-score <-3.0.
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Ready-to-use Therapeutic Food and Hydroxyurea | Ready-to-use Therapeutic Food Alone | Siblings Without SCD
Number analyzed (Participants) | 54 | 54 | 22
percentage of participants | 66.7 | 55.6 | 30.1

ADVERSE EVENTS:
Time Frame: The adverse event data was collected during the participant's 12-week study period, about 7 months after enrollment.
Description: The feasibility trial's primary objectives are to evaluate the intervention's feasibility and safety in children with sickle cell anemia. We, therefore, did not include the outcomes for the siblings in the main results.
Groups:
- Ready-to-use Therapeutic Food and Hydroxyurea: 50 children (5-12 years old) with SCA and severe malnutrition will be randomly allocated to receive Ready-to-use therapeutic food and hydroxyurea (20mg/kg/day)
  hydroxyurea (20mg/kg/day): Treatment of severe malnutrition in children with SCA in northern Nigeria
  Ready-to-use therapeutic food: Treatment of severe malnutrition in children with SCA in northern Nigeria with an additional 500-1000 calories from ready-to-use-therapeutic food
- Ready-to-use Therapeutic Food Alone: 50 children (5-12 years old) with SCA and severe malnutrition will be randomly allocated to receive Ready-to-use therapeutic food alone
  Ready-to-use therapeutic food: Treatment of severe malnutrition in children with SCA in northern Nigeria with an additional 500-1000 calories from ready-to-use-therapeutic food
Arm/Group | Ready-to-use Therapeutic Food and Hydroxyurea | Ready-to-use Therapeutic Food Alone | Siblings Without SCD
All-Cause Mortality (participants affected / at risk) | 1/56 | 0/54 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/56 | 0/54 | 0/22
Other Adverse Events (participants affected / at risk) | 2/56 | 4/54 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ready-to-use Therapeutic Food and Hydroxyurea (N=56) | Ready-to-use Therapeutic Food Alone (N=54) | Siblings Without SCD (N=22)
Prolonged hospitalization (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | NA — One hospitalization was prolonged and met the criteria for an SAE but was deemed unrelated to the study treatment.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ready-to-use Therapeutic Food and Hydroxyurea (N=56) | Ready-to-use Therapeutic Food Alone (N=54) | Siblings Without SCD (N=22)
Pain (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | NA
Acute Chest Syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | NA
Fever (General disorders) | 2 (2) | 3 (3) | NA
Elective Surgery (Ear and labyrinth disorders) | 0 (0) | 1 (1) | NA — Tonsillectomy and Adenoidectomy
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | NA
Malaria (Infections and infestations) | 2 (2) | 3 (3) | NA

LIMITATIONS AND CAVEATS:
The sample size for this feasibility study was not determined with the goal of assessing differences in efficacy between the treatment arms. As a feasibility study, the sample size was not based on determining the difference in efficacy of the 2 treatment arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT03634488/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT03634488/SAP_001.pdf